CLINICAL TRIAL: NCT06357494
Title: Assessment of Thyroid Doppler Ultrasound in Relation to Clinical and Laboratory Parameters in Follow up of Pediatric Graves' Disease
Brief Title: Assessment of Thyroid Doppler Ultrasound in Followup of Pediatric Graves' Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, A.L.Mohamed, Assistant lecturer of pediatrics, Assiut University
Other Study IDs: Thyroid Doppler in Graves'
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Graves' Disease
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All cases of the study will be diagnosed as Graves' by History, examination, laboratory (FT3, FT4, TSH & TRAbs), X-ray on left wrist for bone age, neck grey scale ultrasonography for thyroid gland size, shape, echotexture, vascularity and nodule characters if present with TIRAD score calculation.

Then Color flow doppler ultrasound will be done to asses thyroid volume, number of vessels per square cm and inferior thyroid artery peak systolic velocity, end diastolic velocity and resistive index. Patients then will receive carbimazole antithyroid drug at dose 0.25-0.5 mg/kg/day PO & the dose will be titrated according to thyroid function test after 4-6 weeks.

Beta-adrenergic blockade will be added to all symptomatic cases. Regular follow up will be done every month of first 3 months of diagnosis and then every 3 months for 2 years by clinical and thyroid function test to asses response, compliance, complications, drug side effects, remission and relapses.

Doppler ultrasound will be done at 0, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* All newly diagnosed children with clinical and laboratory hyperthyroidism (high T4 & low TSH) with positive TRAbs.

Exclusion Criteria:

* Patients receiving radioiodine Patients underwent thyroid surgery History of neck radiation or neck surgery

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children who will come at pediatric endocrinology outpatient clinic of Assiut University Children's Hospital meeting our inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-08-05 (Estimated); Primary Completion 2027-04-05 (Estimated); Study Completion 2028-04-05 (Estimated)

PRIMARY OUTCOMES:
thyroid volume | 3 years
number of vessels per square cm of thyroid gland | 2 years
inferior thyroid artery peak systolic velocity | 2 years
end diastolic velocity | 2 years
resistive index | 2 years